CLINICAL TRIAL: NCT00937274
Title: Randomized, Double Blind Placebo-controlled Studies to Evaluate the Effect of an Orally-fed Escherichia Coli (E. Coli) Phage in the Management of ETEC and EPEC Induced Diarrhea in Children
Brief Title: Antibacterial Treatment Against Diarrhea in Oral Rehydration Solution
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08.11.INF
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Diarrhea
Keywords: ETEC EPEC diarrhoea; phage therapy; ORS
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test product (Experimental)
  Interventions: Other: T4 phage cocktail test
- Commercial product (Active Comparator)
  Interventions: Other: Commercial T4 phage cocktail
- Standard care (Placebo Comparator)
  Interventions: Other: standard oral rehydration solution (ORS)

INTERVENTIONS:
Other: T4 phage cocktail test — T4 phages 106 PFU/ ml up to 5 days
  Arms: Test product
Other: Commercial T4 phage cocktail — Treatment as recommended by the manufacturer (Microgen phages)
  Arms: Commercial product
Other: standard oral rehydration solution (ORS) — Standard hospital treatment with ORS
  Arms: Standard care

SUMMARY:
This study hopes to demonstrate the potentials of a new form of therapy for childhood diarrhea, a major cause of morbidity and deaths in Bangladesh and other developing countries, and thus a priority for improving child health.

DETAILED DESCRIPTION:
This randomized double-blind, placebo controlled trial (RCT) aims to evaluate the effect of oral administered E. coli phage in children aged 4-60 months of age with proven ETEC and EPEC diarrhea. Children will be screened to exclude V. cholerae infections by dark field microscopy, rotavirus by stool ELISA, and invasive diarrhoea clinically as well as by stool microscopy, to identify children with possible ETEC and EPEC diarrhoea. Enrolled children will be randomly assigned, in equal numbers, to receive either: (i) a new T4 phage cocktail or (ii) Russian anti-E. coli phage cocktail (Microgen) at the dose recommended by the manufacturer or (iii) only oral rehydration solution (placebo) for 5 days in addition to management of dehydration and continued feeding in accordance with WHO guidelines. Duration of diarrhea, daily and cumulative stool output, volume of oral rehydration solution intake, stool frequency, time to recovery and weight gain will be the main outcome measures. As the dose of phage we intend to use in this therapeutic trial is higher than the dose administered to young children in earlier safety trial, we plan to initially conduct a safety study with these three study products in 45 children with non cholera, non rotavirus and non invasive diarrhea, to randomize equally in the three intervention groups, as for the final study mentioned above. The outcome measures in this safety part will include assessment of laboratory parameters including renal and liver function tests, haematological indices, and microbiological efficacy of phage by measuring phage and E. coli titre in daily stool samples. If the higher dose is found safe, tolerable, and not associated with any significant adverse event, we will proceed to the clinical efficacy trial.

We believe if T4 coli phage is assessed to be effective in the overall diarrhea management, this might lead to development of an affordable and sustainable adjunct to the currently available case management of E. coli diarrhea, benefiting millions of children worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male
2. Age: 6 - 24 months
3. Better nourished (weight for age > 60 NCHS median)
4. H/o. diarrhea of less than 48 hours
5. Written informed consent from either parents/guardian (thumb impression for those who are not literate) for children
6. Negative test results for dark field microscopy of Vibrio cholerae and ELISA test for rotavirus in initial stool samples

Exclusion Criteria:

1. Systemic infection requiring antibiotic treatment
2. Severe malnutrition (W/A < 60%)
3. Unwilling to comply with study procedures
4. Currently participating or have participated in another clinical trial within the last 4 weeks at screening
5. Clinically significant abnormalities from medical history, physical examination, vital signs, haematology, clinical chemistry results, or other laboratory abnormalities
6. Clinically suggestive of invasive diarrhea

Ages: 6 Months to 24 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Assessment of safety, tolerability and efficacy (reduce severity of diarrhea assessed by reduced stool volume and stool frequency) of oral administration of T4 phages in young children with diarrhea due to ETEC and/or EPEC infections | 5 days

SECONDARY OUTCOMES:
Clinical assessment, blood tests, morbidity, duration of hospitalization | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Shafiqul A Sarker, MD, PhD, Principal Investigator — Clinical Sciences Division, ICDDR,B, Mohakhali, Dhaka 1212, Bangladesh
Locations (1):
- Clinical Sciences Division, ICDDR,B, Mohakhali,, Dhaka, Bangladesh

REFERENCES:
- [Derived] Sarker SA, Sultana S, Reuteler G, Moine D, Descombes P, Charton F, Bourdin G, McCallin S, Ngom-Bru C, Neville T, Akter M, Huq S, Qadri F, Talukdar K, Kassam M, Delley M, Loiseau C, Deng Y, El Aidy S, Berger B, Brussow H. Oral Phage Therapy of Acute Bacterial Diarrhea With Two Coliphage Preparations: A Randomized Trial in Children From Bangladesh. EBioMedicine. 2016 Jan 5;4:124-37. doi: 10.1016/j.ebiom.2015.12.023. eCollection 2016 Feb. PMID 26981577